CLINICAL TRIAL: NCT00521404
Title: Phase 2 Multicenter, Open-Label Study of CS-1008, A Humanized Monoclonal Antibody Targeting Death Receptor 5 (DR5), In Combination With Gemcitabine in Chemotherapy Naive Subjects With Unresectable or Metastatic Pancreatic Cancer
Brief Title: Open-label Study of CS-1008 for Subjects With Untreated and Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1008-A-U201
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; chemotherapy naive; unresectable or metastatic pancreatic cancer; CS1008; Gemcitabine; Gemzar
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — tigatuzumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CS-1008 + gemcitabine (Experimental): CS-1008 + gemcitabine
  Interventions: Drug: CS-1008 (humanized anti-DR5 antibody); Drug: gemcitabine

INTERVENTIONS:
Drug: CS-1008 (humanized anti-DR5 antibody) — CS-1008: 8mg/kg loading dose followed by 3mg/kg weekly.
  Other Names: CS1008
Drug: gemcitabine — Gemcitabine - 1000mg/meter sq
  Other Names: Gemzar

SUMMARY:
Phase 2 study to determine the efficacy and safety of CS-1008 when given with gemcitabine to subjects with previously untreated and unresectable (unable to be surgically removed) or metastatic (spread to other areas beyond the pancreas) pancreatic cancer.

DETAILED DESCRIPTION:
Primary Objective:

- To evaluate the efficacy of CS-1008 administered in combination with gemcitabine to chemotherapy naive subjects with unresectable or metastatic pancreatic cancer, based on the progression-free survival at 16 weeks.

Secondary Objectives:

* To evaluate the efficacy of CS-1008 administered in combination with gemcitabine on overall progression-free survival rate, objective response rate, duration of response, and overall survival.
* To determine the pharmacokinetics of BIP CS-1008 and DSC CS-1008.
* To study potential biomarkers of CS-1008 activity
* To assess possible human anti-human antibody formation after exposure to CS-1008
* To evaluate the safety profile of CS-1008 when administered in combination with gemcitabine to chemotherapy naive subjects with unresectable or metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed resectable or metastatic pancreatic cancer; not previously treated with chemotherapy; measurable disease; 18 years of age or older

Exclusion Criteria:

* Anticipation of need for major surgery or radiation therapy during the study
* Heart Disease exclusions: myocardial infarction or unstable angina within the past 6 months; severe or unstable angina pectoris within the past 6 months; coronary or peripheral artery bypass graft within the past 6 mo., etc.
* Clinically significant active infection or history of HIV
* Partial or complete bowel obstruction
* Poorly controlled psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-08-15 (Actual); Primary Completion 2010-08-20 (Actual); Study Completion 2010-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (12):
- United States (12):
  - Birmingham, Alabama
  - Washington D.C., District of Columbia
  - Fort Myers, Florida
  - Atlanta, Georgia
  - Georgia Cancer Specialists, Tucker, Georgia
  - Decatur, Illinois
  - Minneapolis, Minnesota
  - Cincinnati, Ohio
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Temple, Texas
  - Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 65 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at 12 clinic sites in the United States of America. Three (3) of the participants were not treated with the study drug. The data on the 62 treated participants are presented in this report.
Pre-assignment Details: Three participants were enrolled but later failed entry criteria. They did not receive treatment and were not included in this analysis.
Groups:
- CS-1008 + Gemcitabine: Chemotherapy-naïve participants with unresectable or metastatic pancreatic cancer who were administered CS-1008 once weekly without rest, and Gemcitabine once weekly for 3 weeks followed by 1 week of rest. CS-1008 was administered first. Gemcitabine was then administered immediately after completion of the CS-1008 infusion.
Period: Overall Study
Arm/Group | CS-1008 + Gemcitabine
Started | 62
Completed | 0
Not Completed | 62
Not completed — Adverse Event | 13
Not completed — Disease Progression | 33
Not completed — Investigator decision | 5
Not completed — Withdrawal of consent | 3
Not completed — Noncompliance or lack of cooperation | 1
Not completed — Other | 7

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all subjects who received any amount of study drug infusion (ie, CS-1008 or gemcitabine). This analysis set was used to summarize safety variables.
Arm/Group | CS-1008 + Gemcitabine
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 59
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival Rate at 16 Weeks Following Treatment With CS-1008 in Combination With Gemcitabine in Chemotherapy-Naïve Participants With Unresectable or Metastatic Pancreatic Cancer
Description: Progression-free survival rate (PFS) was defined as the time from the date of the first administration of the study drug (Day 1) to the date of the first objective documentation of disease progression or death resulting from any cause, whichever came first at 16 weeks post-treatment with CS-1008.
Time Frame: Baseline to the date of disease progression or death due to any cause (whichever occurs first), up to 16 weeks post dose.
Population: The progression-free survival rate was assessed in the Per-Protocol Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CS-1008 + Gemcitabine
Number analyzed (Participants) | 61
Percentage of participants | 52.5 [39.3 to 64.1]

2. Secondary Outcome: Kaplan-Meier (Non-Parametric) Analysis of Progression-Free Survival Following Treatment With CS-1008 in Combination With Gemcitabine in Chemotherapy-Naïve Participants With Unresectable or Metastatic Pancreatic Cancer
Description: PFS (Progression-free survival) was defined as the time from the date of the first administration of study drug (Day 1) to the date of the first objective documentation of disease progression or death resulting from any cause, whichever came first.
Time Frame: Baseline up to date of disease progression or death due to any cause (whichever occurs first), up to approximately 36 months post dose.
Population: Progression-free survival was assessed in the Per-Protocol Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CS-1008 + Gemcitabine
Number analyzed (Participants) | 61
Percentage of participants
  PFS Rate at 3 Months (%) | 59.0 [45.7 to 70.1]
  PFS Rate at 6 Months (%) | 34.4 [22.9 to 46.3]
  PFS Rate at 9 Months (%) | 21.3 [12.1 to 32.2]
  PFS Rate at 1 Year (%) | 13.1 [6.1 to 22.8]

3. Secondary Outcome: Overall Survival Following Treatment With CS-1008 in Combination With Gemcitabine in Chemotherapy-Naïve Participants With Unresectable or Metastatic Pancreatic Cancer
Description: OS (Overall Survival) was defined as the time from the date of the first administration of study drug (Day 1) to the date of death. If there was no death reported for a subject before the cut-off date for overall survival analysis, overall survival was censored at the last contact date at which the subject was known to be alive.
Time Frame: Baseline to death due to any cause, up to approximately 36 months post dose.
Population: Overall survival was assessed in the Per-Protocol Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CS-1008 + Gemcitabine
Number analyzed (Participants) | 61
Percentage of participants
  OS Rate at 6 Months (%) | 55.7 [42.4 to 67.1]
  OS Rate at 9 Months (%) | 41.0 [28.6 to 52.9]
  OS Rate at 1 Year (%) | 24.6 [14.7 to 35.9]
  OS Rate at 15 Months (%) | 13.1 [6.1 to 22.8]

4. Secondary Outcome: Best Overall Tumor Response Following Treatment With CS-1008 in Combination With Gemcitabine in Chemotherapy-Naïve Participants With Unresectable or Metastatic Pancreatic Cancer
Description: The best overall response the best response (in the order of confirmed complete response [CR], confirmed partial response [PR], unconfirmed CR, unconfirmed PR, stable disease [SD], and progressive disease[PD]) among all overall responses recorded from the start of treatment until the subject withdrew from the study. If there was no tumor assessment after the first infusion of study drug and no clinical disease progression recorded, the best overall response was classified as Unknown. CR was defined as the disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, PD was defined as at least a 20% increase in the sum of diameters of target lesions, and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease PD according to RECIST guideline (version 1.1).
Time Frame: Baseline to up to date of first documented objective response or disease progression (whichever occurs first), up to approximately 36 months post dose.
Population: The best overall tumor response was assessed in the Per-Protocol Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-1008 + Gemcitabine
Number analyzed (Participants) | 61
Participants
  Confirmed CR | 0
  Confirmed PR | 5
  Objective Response (confirmed CR or PR) | 5
  Unconfirmed CR | 0
  Unconfirmed PR | 3
  Stable Disease (SD) | 28
  Progressive Disease (PD) | 14
  Unknown | 11

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events Considered by the Investigator at Least Possibly Related to CS-1008 Experienced by ≥5% of Participants by System Organ Class and Preferred Term
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event (AE) that: emerges during treatment, having been absent at pre-treatment; or reemerges during treatment, having been present at baseline but stopped prior to treatment or worsens in severity during treatment relative to the pre-treatment state when the AE was continuous. The AEs with an onset date on Day 1 (the date on which the first dose of study medication was administered) were counted as a TEAE. An AE that occurred more than 30 days after the last dose of study medication was not included as a TEAE unless it was considered drug-related. A TEAE was considered related to CS-1008 or gemcitabine if the investigator considered the event as possibly, probably, or definitely related to treatment, or if the investigator's assessment of the relationship was unknown.
Time Frame: Baseline up to 30 days post last dose, up to approximately 36 months post dose.
Population: Treatment-Emergent Adverse Events were assessed in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-1008 + Gemcitabine
Number analyzed (Participants) | 62
Participants
  Any TEAE | 43
  Anemia | 8
  Neutropenia | 4
  Thrombocytopenia | 5
  Abdominal Pain | 5
  Constipation | 8
  Diarrhea | 8
  Nausea | 22
  Vomiting | 8
  Asthenia | 11
  Fatigue | 20
  Oedma peripheral | 12
  Pyrexia | 10
  Haemoglobin decreased | 6
  Neutrophil count decreased | 5
  White blood cell count decreased | 4
  Anorexia | 8
  Dysgeusia | 4
  Headache | 6
  Rash | 4
  Hypertension | 4

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events Considered by the Investigator at Least Possibly Related to Gemcitabine Experienced by ≥5% of Participants by System Organ Class and Preferred Term
Description: as for outcome 5
Time Frame: Baseline up to 30 days post last dose, up to approximately 36 months post dose.
Population: Treatment-emergent adverse event was assessed in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-1008 + Gemcitabine
Number analyzed (Participants) | 62
Participants
  Any TEAE | 54
  Anemia | 15
  Leukopenia | 4
  Lymphopena | 5
  Thrombocytopenia | 11
  Abdominal distension | 4
  Abdominal pain | 5
  Constipation | 7
  Diarrhea | 11
  Nausea | 31
  Vomiting | 20
  Asthenia | 12
  Chills | 5
  Fatigue | 22
  Oedema peripheral | 10
  Pyrexia | 11
  Haemoglobin decreased | 10
  Neutrophil count decreased | 9
  Platelet count decreased | 9
  White blood cell count decreased | 7
  Anorexia | 8
  Dehydration | 5
  Dysgeusia | 4
  Headache | 6
  Alopecia | 4
  Night Sweats | 4
  Rash | 5

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected and reported from when the first dose of study drug was administered to 30 days after the last dose of study drug. Treatment-emergent AE (TEAE) and serious AE data were collected from baseline up to 36 months postdose.
Description: A treatment-emergent AE (TEAE) was defined as an AE that emerges during treatment, having been absent at pre-treatment; or reemerges during treatment, having been present at baseline but stopped prior to treatment; or worsens in severity during treatment after initiating the study drug until 30 days after last dose of the study drug, unless it was considered drug related.
Arm/Group | CS-1008 + Gemcitabine
All-Cause Mortality (participants affected / at risk) | 61/62
Serious Adverse Events (participants affected / at risk) | 35/62
Other Adverse Events (participants affected / at risk) | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CS-1008 + Gemcitabine (N=62)
Anaemia (Blood and lymphatic system disorders) | 4
Atrial fibrillation (Cardiac disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Disease Progression (General disorders) | 2
Pyrexia (General disorders) | 2
Cholangitis (Hepatobiliary disorders) | 2
Clostridium difficile colitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Cerebral infarction (Nervous system disorders) | 1
Confusional State (Psychiatric disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CS-1008 + Gemcitabine (N=62)
Anaemia (Blood and lymphatic system disorders) | 21
Leukopenia (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 14
Tachycardia (Cardiac disorders) | 5
Visual impairment (Eye disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 32
Abdominal pain upper (Gastrointestinal disorders) | 8
Ascites (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 31
Diarrhea (Gastrointestinal disorders) | 24
Dry Mouth (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 12
Dysphagia (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 47
Oral pain (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 34
Asthenia (General disorders) | 17
Chest discomfort (General disorders) | 4
Chest pain (General disorders) | 4
Chills (General disorders) | 10
Fatigue (General disorders) | 43
Malaise (General disorders) | 4
Mucosal inflammation (General disorders) | 4
Oedema (General disorders) | 4
Oedema Peripheral (General disorders) | 25
Pain (General disorders) | 9
Pyrexia (General disorders) | 30
Jaundice (Hepatobiliary disorders) | 4
Pneumonia (Infections and infestations) | 5
Sinusitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 7
Procedural pain (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 5
Gamma-glutamyltranferase increased (Investigations) | 4
Haemoglobin decreased (Investigations) | 10
Neutrophil count decreased (Investigations) | 9
Platelet count decreased (Investigations) | 9
Weight decreased (Investigations) | 13
Weight increased (Investigations) | 4
White blood cell count decrased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 22
Dehydration (Metabolism and nutrition disorders) | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Hyponatraemia (Metabolism and nutrition disorders) | 10
Artralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 15
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 14
Neuropathy peripheral (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 18
Depression (Psychiatric disorders) | 10
Insomnia (Psychiatric disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Rales (Respiratory, thoracic and mediastinal disorders) | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6
Night sweats (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 9
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No